CLINICAL TRIAL: NCT01799629
Title: Efficacy of Prophylactic Glycerin Suppositories for Feeding Intolerance in Very Low Birth Weight Preterm Infants: a Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issue
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Dr. Sulaiman Alhabib Medical City, Riyadh (Other); Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohammad Khadawardi, Consultant Neonatology, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2121 110
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Glycerin suppositories; Feeding intolerance; preterm infants; prophylactic use; elimination of meconium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive the glycerin suppository
  Interventions: Drug: Glycerin suppositories
- Control (No Intervention): Normal care

INTERVENTIONS:
Drug: Glycerin suppositories
  Arms: Intervention

SUMMARY:
To evaluate the efficacy of prophylactic glycerin suppositories will accelerate the elimination of meconium from the large intestine and thus reduce the incidence of feeding intolerance in very low birth weight (VLBW) infants

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with birth weight < 1250g.
2. Inborn or outborn infants
3. Less than 72 hours of age.

Exclusion Criteria:

1. Congenital malformations.
2. Acute abdomen needing surgical intervention.
3. Severity of illness such that death is likely in the first few days after birth.
4. Inability to get the parental consent.

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
days to achieve full tolerated feeding (breast milk or formula) by NGT or by mouth (140cc/kg/day) | 2years

SECONDARY OUTCOMES:
Incidence of feeding intolerance | 2years
  which is defined by the presence of GRVs > 50 % of the previous feed for two consecutive feeds in addition to two of the following: I. Abdominal distention > 1 cm in 12 hour. II. Abdominal tenderness. III. Vomiting. IV. Bile stained aspirate.
Incidence of necrotizing enterocolitis (NEC) | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Emad M Khadawardi, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (3):
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & Research Centre, Riyadh
  - Security Forces Hospital, Riyadh
  - Sulaiman Al habib Medical Center, Riyadh